CLINICAL TRIAL: NCT03392701
Title: Possible Links Between Inflammation and Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barmherzige Brüder Linz (Other)
Responsible Party: Principal Investigator, Martin Clodi, Prim. Univ.-Prof. Dr. Martin Clodi, Head of Internal Medicine,, Barmherzige Brüder Linz
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LPS lipid metabolism
Record Dates: First submitted 2017-12-21; First posted 2018-01-08 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Sepsis; Inflammation; LPS; Lipid Metabolism Disorder
MeSH Terms: conditions — Sepsis; Inflammation; Lipid Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LPS infusion (Experimental): infusion of LPS 2 ng/kg over 5 minutes
  Interventions: Biological: LPS infusion
- Placebo (Placebo Comparator): NaCl
  Interventions: Biological: LPS infusion

INTERVENTIONS:
Biological: LPS infusion — infusion of LPS 2 ng/kg over 5 minutes

SUMMARY:
It has been recognized lately that sepsis and inflammation has an important impact on lipid metabolism and that the extent of hypocholesterolemia may even be a marker of severity of illness. However, the interplay between inflammation and the marked changes in lipid metabolism remain to be sufficiently understood. Importantly, the exact kinetics of lipid parameters in inflammatory conditions are yet to be explored. This study aims to investigate the interaction between inflammation and lipid metabolism using the human endotoxin model (LPS infusion) in ten healthy volunteers in a single blinded randomized placebo controlled cross-over design.

DETAILED DESCRIPTION:
Sepsis is a severe clinical syndrome with still limited means of therapy and often poor prognosis. It has been recognized lately that sepsis and inflammation has an important impact on lipid metabolism and that the extent of hypocholesterolemia may even be a marker of severity of illness.

This study aims to investigate the interaction between inflammation and lipid metabolism and the possible role of various markers of lipid metabolism including apolipoprotein B, apoA1 and lipoprotein(A) using the human endotoxin model in ten healthy volunteers. In this model, volunteers are infused intravenously with bacterial lipopolysaccharide (LPS, 2 ng/kg over 5 minutes) to simulate human sepsis. Immediately after the infusion of LPS, proinflammatory cytokines and other mediators are elevated just as they are in common sepsis. This widely used model thus represents a reliable method for evaluating conditions during inflammation.

In this study, LPS will be administered to ten healthy male volunteers aged 18-40 years and plasma levels of lipid parameters including those described above will subsequently be measured repeatedly to evaluate the influence of LPS on lipid metabolism and detailed kinetics of lipid parameters.

This project is planned as a prospective, single blinded randomized, placebo controlled cross-over study. Participants must be free of disease history and previous anaphylactic events, must not be on any medication and will be screened for medical disorders including renal, hepatic and cardiovascular conditions, thrombophilia and infections in an initial medical examination. Each participant will be studied on two different study days with a washout period of at least 14 days, on which either LPS (National Reference Bacterial Endotoxin, lot EC-6, prepared from Escherichia coli 0113, USPC, Inc. Rockville, MD) and saline or saline alone as a placebo will be administered. LPS will be infused in a dosage of 2 ng/kg over a period of 5 minutes. Participants will be studied after an overnight fast and after 24 hours without smoking and without consumption of caffeine-containing beverages in order to ensure standard baseline conditions. During the study, subjects will rest in a supine position. Infusion and sampling will be done using two separate intravenous catheters.

Blood samples will be centrifuged, transferred into chilled tubes and placed on ice. Plasma will be frozen at -80°C until it will be assayed. Plasma and urine sodium, potassium, creatinine and glucose will be measured via routine laboratory techniques.

A case record form will be completed for each volunteer and data will subsequently be handled in an anonymous manner. Data will be analysed using repeated measures ANOVA.

In summary, this study aims to evaluate the interactions between sepsis and lipid metabolism using the human endotoxin model. Such knowledge could improve the understanding of the pathophysiology in sepsis and may lead to the development of novel therapeutic strategies. Insights on possible interactions between inflammation and lipid metabolism could also enlighten pathophysiological pathways in metabolic syndrome and type 2 diabetes mellitus causing chronic low-grade inflammation with potential impact on various medical fields.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 40 years
* Written informed consent
* No disease history
* non-smoker
* BNP level within the normal range
* Normal renal function (serum creatinine of 1.3 mg/dL and/or creatinine clearance greater than 80ml/min)

Exclusion Criteria:

* Systolic blood pressure < 90 mmHg
* Subjects on any medication
* History of anaphylaxis
* Probands who suffer from infectious disease

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male
Enrollment: 10 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
lipid kinetics | 48 hours
  levels of lipid parameters including LDL, HDL, lipoprotein(a), apolipoprotein A1 and apoB will be measured at multiple timepoints (t0, t15, t30, t60, t120, t180, t360, 24h and 48h) in order to evaluate the detaile kinetics of lipid parameters in inflammatory condidtions

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Heinzl, MD, Study Chair — Barmherzige Brüder Linz
Locations (1):
- Barmherzige Brüder Linz - Innere Medizin, Linz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Heinzl MW, Resl M, Klammer C, Fellinger P, Schinagl L, Obendorf F, Feldbauer R, Pohlhammer J, Wagner T, Egger M, Dieplinger B, Clodi M. SUBCLINICAL KIDNEY INJURY IS CAUSED BY A MODERATE SINGLE INFLAMMATORY EVENT. Shock. 2022 Jul 1;58(1):14-19. doi: 10.1097/SHK.0000000000001942. Epub 2022 Jul 19. PMID 35616594
- [Derived] Millischer V, Heinzl M, Faka A, Resl M, Trepci A, Klammer C, Egger M, Dieplinger B, Clodi M, Schwieler L. Intravenous administration of LPS activates the kynurenine pathway in healthy male human subjects: a prospective placebo-controlled cross-over trial. J Neuroinflammation. 2021 Jul 17;18(1):158. doi: 10.1186/s12974-021-02196-x. PMID 34273987
- [Derived] Heinzl MW, Resl M, Klammer C, Egger M, Dieplinger B, Clodi M. Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Is Not Induced in Artificial Human Inflammation and Is Not Correlated with Inflammatory Response. Infect Immun. 2020 Feb 20;88(3):e00842-19. doi: 10.1128/IAI.00842-19. Print 2020 Feb 20. PMID 31843964